CLINICAL TRIAL: NCT06810466
Title: A Single-blind, Parallel-group, Randomized, Placebo-controlled Clinical Trial, to Evaluate the Effects of Two Different Formulations of a Dietary Supplement on the Lipid Profile in Subjects with Mild Hypercholesterolemia
Brief Title: Evaluation of the Effects of Two Dietary Supplement Formulations on the Lipid Profile in Mild Hypercholesterolemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Informapro Srl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COLE_TRIAL_2023; COLE_TRIAL_2023 (Other: IBSA Farmaceutici Italia Srl)
Record Dates: First submitted 2025-01-08; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Hypercholesterolemia and Hyperlipidemia; Supplementation
Keywords: mild hypercholesterolemia; supplement; lipid profile; dietary supplement
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized, placebo-controlled clinical trial, followed by an open label phase
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Product A (Experimental): Innovative formulation of dietary supplement
  Interventions: Dietary Supplement: Test Product A
- Test Product B (Active Comparator): Classic formulation of dietary supplement
  Interventions: Dietary Supplement: Test Product B
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Test Product A — Innovative formulation of a dietary supplement for mild hypercholesterolemia. Test Product A will be admistered daily for 8 weeks. After the fist 8 weeks, this arm will continue with the intake of the Product Test A for other 8 weeks.
  Arms: Test Product A
Dietary Supplement: Test Product B — Classic formulation of a dietary supplement for mild hypercholesterolemia. After the fist 8 weeks, this arm will continue with the intake of the Product Test A for other 8 weeks.
  Arms: Test Product B
Dietary Supplement: Placebo — Placebo does not contain functional components and is indistinguishable from Product Test B.
  After the fist 8 weeks, this arm will continue with the intake of the Product Test A for other 8 weeks.
  Arms: Placebo

SUMMARY:
A single-center, randomized, parallel-group, double-blind, placebo-controlled clinical study followed by an open-label phase to evaluate the effects of a new formulation of a supplement on lipid profile in subjects with mild hypercholesterolemia who are non-responsive to the Mediterranean diet.

The study population consists of 99 subjects with mild hypercholesterolemia who are non-responsive to the Mediterranean diet. The participants will be divided into three groups:

Group A: Test Product A (study product) Group B: Test Product B (comparative product) Placebo group: placebo

The following visits are scheduled during the study:

T-2 (day -35) - Screening visit, 5 weeks before T0 T-1 (day -28) - Enrollment visit, 4 weeks before T0 T0 (day 0) - Randomization visit, baseline T1 (day 56) - Interim visit, 8 weeks after T0 T2 (day 112) - Final visit, 16 weeks after T0 After the first 8 weeks of the study (double-blind), all three groups will continue with only Product A for an additional 8 weeks. This experimental design aims to highlight whether any differences between Test Product A and Test Product B observed during the first 8 weeks can be minimized when both arms receive the same treatment. Additionally, the effect of Product A will be observed at 8 and 16 weeks, thus providing efficacy data over a longer treatment period. This may also provide insights into the potential achievement of a plateau. Regarding the placebo group, it will be possible to distinguish the effect of the diet alone from the combined effect of the diet and supplementation with Test Product A.

ELIGIBILITY:
Inclusion Criteria:

* Prevention of cardiovascular disease
* Low cardiovascular risk (< 5%)
* Sub-optimal serum levels of LDL-C (130-136 mg/dl; 3.37-4.14 mmol/l) and/or non-HDL-C (160-190 mg/dl; 4.14-4.92 mmol/l) at T-2
* Signature of informed consent.

Exclusion Criteria:

* Patients with cardiovascular disease (in secondary prevention) or at risk of cardiovascular disease after 10 years (cardiovascular risk >/= 5)
* diabetes mellitus
* Taking hypolipemiants, supplements or drugs that may involve lipid metabolism
* Hypertension treatment not stabilized for at least 3 months
* History of ongoing kidney, thyroid, gastrointestinal, muscle or liver disease
* Any medical-surgical treatment that may limit adherence to the study protocol
* Pregnant and/or breastfeeding women

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Low-Density Lipoprotein Cholesterol (LDL-C) Serum Concentration After Target Product A Treatment | At baseline (T0) and at 8 weeks.
  Evaluation of absolute value change in Low-Density Lipoprotein Cholesterol (LDL-C) serum concentration (expressed as mg/dL), at 8 weeks (T1) of dietary supplementation with Test Product A vs baseline (T0).
Low-Density Lipoprotein Cholesterol (LDL-C) Serum Concentration After Target Product A Treatment | At baseline (T0) and at 8 weeks.
  Evaluation of the percentage variation (%) in Low-Density Lipoprotein Cholesterol (LDL-C) serum concentration at 8 weeks (T1) of dietary supplementation with Test Product A, compared to baseline (T0).

SECONDARY OUTCOMES:
Low-Density Lipoprotein Cholesterol (LDL-C) Serum Concentration After Treatment with Target Product B | At baseline (T0) and at 8 weeks.
  Evaluation of absolute value change in Low-Density Lipoprotein Cholesterol (LDL-C) serum concentration (expressed as mg/dL), at 8 weeks (T1) of dietary supplementation with Test Product B vs baseline (T0).
Low-Density Lipoprotein Cholesterol (LDL-C) Serum Concentration After Treatment with Target Product B | At baseline (T0), and at 8 weeks (T1)
  Evaluation of the percentage change (%) in Low-Density Lipoprotein Cholesterol (LDL-C) serum concentration at 8 weeks (T1) of dietary supplementation with Test Product B, compared to baseline (T0)
Serum Total Cholesterol Concentration (TC) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Serum Total Cholesterol concentration (TC; expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Serum Total Cholesterol Concentration (TC) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Serum Total Cholesterol concentration (TC) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Low-Density Lipoprotein Cholesterol (LDL-C) Serum Concentration | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in serum concentrations of Low-Density Lipoprotein Cholesterol (LDL-C; expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Low-Density Lipoprotein Cholesterol (LDL-C) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Low-Density Lipoprotein Cholesterol (LDL-C) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
High-Density Lipoprotein Cholesterol (HDL-C) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in serum concentrations of High-Density Lipoprotein Cholesterol (HDL-C; expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
High-Density Lipoprotein Cholesterol (HDL-C) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in serum concentrations of High-Density Lipoprotein Cholesterol (HDL-C) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Non High-Density Lipoprotein Cholesterol (Non-HDL-C) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in serum concentrations of Non High-Density Lipoprotein Cholesterol (Non-HDL-C; expressed in mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Non High-Density Lipoprotein Cholesterol (Non-HDL-C) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in serum concentrations of Non High-Density Lipoprotein Cholesterol (Non-HDL-C) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Triglycerides (TG) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of absolute value change in Triglycerides (TG) serum concentration (expressed as mg/dL), at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Triglycerides (TG) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in serum concentrations of Triglycerides (TG) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Apolipoprotein B | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in serum concentrations of Apolipoprotein B (expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0)
Apolipoprotein B | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in serum concentrations of Apolipoprotein B at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Systolic Blood Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Systolic Blood Pressure (expressed as mmHg) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Systolic Blood Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Systolic Blood Pressure at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Diastolic Blood Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Diastolic Blood Pressure (expressed as mmHg) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Diastolic Blood Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Diastolic Blood Pressure at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Mean Arterial Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute change in Mean Arterial Pressure (expressed in mmHg) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Mean Arterial Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Mean Arterial Pressure at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Pulse Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute change in Pulse Pressure (expressed in mmHg) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Pulse Pressure | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Pulse Pressure at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Flow-Mediated Dilation (FMD) - Endothelial Function | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Flow-Mediated Dilation (FMD), measured as the percentage increase in artery diameter during hyperemia, at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0)
Body Weight | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Weight (kg) at 8 weeks (T1) and 16 weeks (T2), compared to baseline (T0), within and between groups.
Body Weight | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) Weight at 8 weeks (T1) and 16 weeks (T2), compared to baseline (T0), within and between groups.
Body Mass Index (BMI) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Body Mass Index (BMI; kg/m²), at 8 weeks (T1) and 16 weeks (T2), compared to baseline (T0), within and between groups.
Body Mass Index (BMI) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Body Mass Index (BMI), at 8 weeks (T1) and 16 weeks (T2), compared to baseline (T0), within and between groups.
Glutamic Oxaloacetic Transaminase (GOT) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Glutamic Oxaloacetic Transaminase (GOT) concentration (expressed as U/L) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Glutamic Oxaloacetic Transaminase (GOT) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Glutamic Oxaloacetic Transaminase concentration (GOT; expressed as U/L) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Gamma-Glutamyl Transferase (Gamma - GT) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Gamma-Glutamyl Transferase (Gamma - GT) concentration (expressed as U/L) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Gamma-Glutamyl Transferase (Gamma - GT) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Gamma-Glutamyl Transferase (Gamma - GT) concentration at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Glutamic Pyruvate Transaminase (GPT) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Glutamic Pyruvate Transaminase (GPT) concentration (expressed as U/L) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Glutamic Pyruvate Transaminase (GPT) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Glutamic Pyruvate Transaminase (GPT) concentration at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Serum Uric Acid | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Serum Uric Acid concentration (expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Serum Uric Acid | At Baseline (T0), at 8 weeks (T1), and at 16 weeks (T2)
  Evaluation of the percentage change (%) in Serum Uric Acid concentrations at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Creatinine Concentration | At Baseline (T0), at 8 weeks (T1), and at 16 weeks (T2).
  Evaluation of the absolute value change in Creatinine Concentration (expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Creatinine Concentration | At baseline (T0), 8 weeks (T1) and 16 weeks (T2).
  Evaluation of the percentage change (%) in Creatinine Concentration at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Creatine phosphokinase (CPK) Concentration | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Creatine Phosphokinase (CPK) concentration (expressed in mcg/L) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline.
Creatine phosphokinase (CPK) Concentration | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Creatine Phosphokinase (CPK) concentration at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline.
Number of subjects with LDL-C normal concentration | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation at 8 weeks (T1) and 16 weeks (T2) of the number of subjects in each group with LDL-C levels (mg/dL) within the normal range of concentration.
Fasting Blood Glucose Concentration | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the absolute value change in Fasting Blood Glucose concentration (expressed as mg/dL) at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Fasting Blood Glucose Concentration | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Evaluation of the percentage change (%) in Fasting Blood Glucose concentration at 8 weeks (T1) and 16 weeks (T2), within and between groups, compared to baseline (T0).
Cardiovascular Risk (CV) | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Assessment of the Cardiovascular Risk (CV), based on Cardiovascular Risk Chart, at 8 weeks (T1) and 16 weeks (T2), compared with baseline (T0).
Patients' compliance with the treatment | At baseline (T0), 8 weeks (T1), and 16 weeks (T2)
  Assessment of patient's compliance with the treatment by calculating the percentage ratio between the number of capsules taken and the number of capsules expected at 8 weeks (T1), and 16 weeks (T2), in each group and intergroup vs baseline (T0).
  Number of patients: 99; assigned treatment: Test Product A; Test product B; Placebo.
Patients' Tolerability of the assigned treatment | At 8 weeks (T1) and at 16 weeks (T2)
  Evaluation of Patients' Tolerability of the assigned treatment using the Visual Analogue Scale (VAS), with scores ranging from 1 to 10, where higher scores indicate greater tolerability, assessed at 8 weeks (T1) and 16 weeks (T2), with intra-group and inter-group evaluations.
  Number of patients: 99; assigned treatments: Test Product A, Test Product B, Placebo.
Patient acceptability of the assigned treatment | At 8 weeks (T1) and at 16 weeks (T2)
  Evaluation of patient acceptability of the assigned treatment using the Visual Analogue Scale (VAS), with scores ranging from 1 to 10, where higher scores indicate greater acceptability, assessed at 8 weeks (T1) and 16 weeks (T2), with intra-group and inter-group evaluations.
  Number of patients: 99; assigned treatments: Test Product A, Test Product B, Placebo.
Patients' adherence to diet | Baseline (T0), 8 weeks (T1), 16 weeks (T2)
  Assessment of patients' adherence to diet based on the food history questionnaire recording at baseline (T0), 8 weeks (T1), 16 weeks (T2), and intra-group and intergroup evaluation.
Implementation of patients' lifestyle | At Baseline (T0), at 8 weeks (T1), and at 16 weeks (T2)
  Measurement of the rate of successful implementation of patients' lifestyle changes, through the evaluation of the prescription of physical exercise (brisk walking or cycling for 20-30 minutes, 3-5 times per week) by the investigator, assessed at baseline (T0), 8 weeks (T1), and 16 weeks (T2), with both intra-group and inter-group evaluations
Monitoring of adverse events | Through study completion, an average of 1 year
  Collection of adverse events after treatment with product A, B and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Results, data, workflows, and tools may be made available through publication, presentations at scientific meetings.